CLINICAL TRIAL: NCT05340491
Title: Chemoradiotherapy Combined With Programmed Death 1 Antibody in Recurrent Nasopharyngeal Carcinoma: A Multicenter, Open-label, Randomised, Controlled, Phase III Trial
Brief Title: Chemoradiotherapy Plus Anti-PD1 in Recurrent NPC: A Multicenter, Open-label, Randomised, Controlled, Phase III Trial
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Sun Yat-sen University (Other)
Responsible Party: Principal Investigator, Zhao Chong, Prof., Sun Yat-sen University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: B2022-111-01
Record Dates: First submitted 2022-04-09; First posted 2022-04-22 (Actual); Last update posted 2022-08-31 (Actual); Status verified 2022-08

CONDITIONS: Nasopharyngeal Carcinoma
Keywords: locoregional relapse; nasopharyngeal carcinoma; chemoradiotherapy; PD-1 antibody; efficacy; toxicity
MeSH Terms: conditions — Nasopharyngeal Carcinoma | interventions — toripalimab; Drug Therapy; Radiotherapy, Intensity-Modulated

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Chemoradiotherapy+anti-PD-1 (Experimental): Patients in this arm will receive three cycles of GP chemotherapy plus PD-1 antibody, then receive IMRT and PD-1 antibody maintenance for eight cycles.
  Interventions: Drug: Toripalimab; Drug: Chemotherapy; Radiation: Intensity modulated radiotherapy
- Chemoradiotherapy (Active Comparator): Patients in this arm will receive three cycles of GP chemotherapy, then receive IMRT.
  Interventions: Drug: Chemotherapy; Radiation: Intensity modulated radiotherapy

INTERVENTIONS:
Drug: Toripalimab — 240mg, D1, every 3 weeks per cycle, three cycles with chemotherapy and eight cycles after IMRT
  Other Names: JS001
  Arms: Chemoradiotherapy+anti-PD-1
Drug: Chemotherapy — Gemcitabine: 1.0g/m2, D1 and D8, Cisplatin 80mg/m2, D1, every 3 weeks per cycle, total three cycles
  Other Names: GP
Radiation: Intensity modulated radiotherapy — total 60-66Gy, 1.8-2.0Gy/f/day
  Other Names: IMRT

SUMMARY:
This is a multicenter, open-label, randomized, controlled, phase III trial. The purpose of this trial is to evaluate the efficacy and toxicity of anti-PD-1 antibody combined with chemoradiotherapy versus chemoradiotherapy alone in recurrent nasopharyngeal carcinoma patients.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed as local with or without regional recurrence after ≥1 year of radical treatment;
* Not suitable for surgery;
* Histologic diagnosis of NPC (WHO II/III);
* TNM stage rII-IVa (AJCC/UICC 8th);
* ECOG 0-1 point;
* No treatment to rNPC prior, such as radiotherapy, chemotherapy, immunotherapy or biotherapy;
* No contraindications to immunotherapy or chemoradiotherapy;
* Adequate marrow function: WBC count ≥ 3×10E9/L, NE count ≥ 1.5×10E9/L, HGB ≥ 90g/L, PLT count ≥ 100×10E9/L;
* Adequate liver function: ALT/AST ≤ 2.5×ULN, TBIL ≤ 2.0×ULN;
* Adequate renal function: BUN/CRE ≤ 1.5×ULN or endogenous creatinine clearance ≥ 60ml/min (Cockcroft-Gault formula);
* Take effective contraceptions during and two months after treatment;
* Patients must be informed of the investigational nature of this study and give written informed consent.

Exclusion Criteria:

* Treated with anti-tumor Chinese medicine treatment;
* Have recurrence with local necrosis;
* Have ≥G3 late toxicities, except for skin, subcutaneous tissue or mucosa;
* Unexplained fever > 38.5, except for tumor fever;
* Treated with ≥ 5 days antibiotics one month before enrollment;
* Have active autoimmune disease (e.g., uveitis, enteritis, hepatitis, hypophysitis, nephritis, vasculitis, hyperthyroidism, and asthma requiring bronchodilator therapy); Have a known history of human immunodeficiency virus (HIV), active Hepatitis B (HBV-DNA ≥10E3copiers/ml) or hepatitis C virus (HCV) antibody positive; Have previously treated with PD-1 antibody or other immunotherapy for PD-1/PD-L1 pathway;
* Have New York Heart Association (NYHA) class 3 or 4, unstable angina, myocardial -infarction within 1 year, or clinically meaningful arrhythmia that requires treatment;
* Have known allergy to large molecule protein products or any compound of study therapy;
* Pregnant or breastfeeding;
* Prior malignancy except adequately treated non-melanoma skin cancer, in situ cervical cancer, and papillary thyroid carcinoma;
* Have received a live vaccine within 30 days of planned start of study therapy Has psychiatric drug or substance abuse disorders that would interfere with cooperation with the requirements of the trial;
* Any other condition, including mental illness or domestic/social factors, deemed by the investigator to be likely to interfere with a patient's ability to sign informed consent, cooperate and participate in the study, or interferes with the interpretation of the results.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 212 (Estimated)
Dates: Start 2022-04-01 (Actual); Primary Completion 2024-12 (Estimated); Study Completion 2027-12 (Estimated)

PRIMARY OUTCOMES:
Overall survival | three years
  Defined as the time from date of recruitment to death from any cause.

SECONDARY OUTCOMES:
Failure-free survival | three years
  Defined as the time from date of recruitment to documented relapse or death from any cause.
Objective response rate through study completion, an average of nine months | through study completion, an average of nine months
  The rate of patients get CR or PR after treatment
Disease control rate through study completion, an average of nine months | through study completion, an average of nine months
  The rate of patients get CR or PR or SD after treatment
Incidence of nasopharyngeal necrosis and hemorrhage up to 3 years | up to three-year follow-up
  Incidence of nasopharyngeal necrosis and hemorrhage after receiving treatment
Acute toxicities were graded using the Common Toxicity Criteria for Adverse Events version 5.0 (CTCAE v5.0) | through study completion, an average of nine months
  Acute toxicities were graded using the Common Toxicity Criteria for Adverse Events version 5.0 (CTCAE v5.0) for chemotherapy and immunotherapy-specific toxicities, and the Radiation Therapy Oncology Group (RTOG) radiation morbidity scoring criteria for radiotherapy-specific toxicities.
Late toxicity | three years
  Late toxicities were assessed annually using the RTOG radiation morbidity scoring criteria.
Quality of life through study completion, up to 3 years | up to three-year follow-up
  Evaluated with questionnaire of EuroQoL 5 dimension, 5 level health state utility index (EQ-5D-5L).

CONTACTS AND LOCATIONS:
Overall Officials: Chong Zhao, MD PhD, Principal Investigator — Sun Yat-sen University
Locations (12):
- China (12):
  - Sun Yat-sen University Cancer Center, Guangzhou, Guangdong
  - Peking University Third Hospital, Beijing
  - Sichuan Cancer Hospital, Chengdu
  - Fujian Province Cancer Hospital, Fuzhou
  - Guizhou Cancer Hospital, Guiyang
  - Zhejiang Cancer Hospital, Hangzhou
  - Jiangxi Cancer Hospital, Nanchang
  - The First Affiliated Hospital of Guangxi Medical University, Nanning
  - Fudan University Shanghai Cancer Center, Shanghai
  - Zhongnan Hospital of Wuhan University, Wuhan
  - Xijing Hospital, Xi'an
  - The First Affiliated Hospital of Xiamen University, Xiamen

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- See also: Home Page of Sun Yat-sen University Cancer Center — http://www.sysucc.org.cn